CLINICAL TRIAL: NCT02581722
Title: A Safety and Efficacy Study of Non-surgical MC Device on PrePex Adolescent Male Population, Including Contraindicated Subjects Scheduled to Undergo Circumcision in an Effort to Prevent the Spread of HIV in Resource Limited Settings
Brief Title: Safety and Efficacy Study of Non-Surgical MC Device for Adolescent Male Population Including Contraindicated Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ministry of Health, Rwanda (Other Government)
Responsible Party: Principal Investigator, Vincent Mutabazi, Director of the Research Grants Unit, Ministry of Health, Rwanda
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RMC-04A
Record Dates: First submitted 2015-10-19; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Circumcision, Adolescents
Keywords: PrePex, Male Circumcision, HIV Prevention, Adolescents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adolescent male population (Experimental): Male circumcision using the PrePex device among healthy adolescent males and contraindicated subjects due to Preputial adhesions and /or narrow foreskin/Phimosis
  Interventions: Device: PrePex Device

INTERVENTIONS:
Device: PrePex Device — The PrePex device is designed to enable conducting male circumcision procedure that is bloodless with no anesthesia and no sutures. For contraindicated subjects, a preparation procedure will take place.

SUMMARY:
A new Male Circumcision (MC) device, PrePex, has shown great promise as a way to radically shift the MC landscape. PrePex is an innovative circumcision device requiring no injected anesthesia, sutures, or sterile settings. Moreover, it is designed for use by minimally skilled healthcare professionals rather than surgeons. Two initial studies conducted in Rwanda in 2010 and 2011 demonstrated an excellent safety profile when the procedure was performed by skilled physicians

DETAILED DESCRIPTION:
Rwanda Has also completed a third study to assess the safety and efficacy of MC when performed by nurses using PrePex in both rural and urban hospitals, Device safety was assessed by the rate of clinical adverse events and device-related incidents attributed to the PrePex device and its procedures, the study report was shared with the WHO Male Circumcision Technical Advisory Group. On February 2011 the WHO provided Rwanda with recommendation to phase in MC scale up with the PrePex device on adults. Moreover the WHO recommended Rwanda to study the PrePex for use on adolescent population, starting on ages 15-17 and thereafter on ages 12-14 and 10-12.

ELIGIBILITY:
Inclusion Criteria:

* Adolescent Males in ages - 10 to 17 years
* Uncircumcised
* Subject wants to be circumcised
* Subject assent to the procedure
* Legal guardian consent to the procedure
* Subject with or without the following conditions: Preputial adhesions and /or narrow foreskin/Phimosis
* Able to understand the study procedures and requirements
* Agrees to abstain from sexual intercourse for 8 weeks after circumcision
* Agrees to abstain from masturbation for at least 2 weeks after Removal
* Agrees to return to the health care facility for follow-up visits (or as instructed) after his circumcision for a period of 7 weeks post removal (8 weeks total)
* Subject able to comprehend and freely give informed consent for participation in this study and is considered by the investigator to have good compliance for the study
* Subject agrees to anonymous video and photographs of the procedure and follow up visits.

Exclusion Criteria:

* Legal guardian withholds consent
* Active genital infection, anatomic abnormality or other condition, which in the opinion of the investigator prevents the subject from undergoing a circumcision
* Subject with the following diseases/conditions: paraphimosis, warts under the prepuce, torn or tight frenulum, hypospadias, epispadias
* Known bleeding / coagulation abnormality, uncontrolled diabetes
* Subject that to the opinion of the investigator is not a good candidate
* Subject does not agree to anonymous video and photographs of the procedure and follow up visits.

Ages: 10 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2015-08; Primary Completion 2015-09 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events on adolescent male population including contraindicated subjects in ages 10 to 17 | up to 7 weeks

SECONDARY OUTCOMES:
Glans fully exposed | Up to 7 weeks
The pain at key time points | Up to 7 weeks
Time to complete healing | Up to 7 weeks
Time to numb the foreskin using topical Lidocaine 5% cream - for contraindicated subjects only | Up to 7 weeks
Rate of side effects | Up to 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Mutabazi, M.D., Principal Investigator — Ministry of Health, Rwanda
Locations (1):
- Rwanda Military Hospital, Kigali, Kigali, Rwanda

REFERENCES:
- See also: Rwanda Biomedical Center — http://www.rbc.gov.rw/